CLINICAL TRIAL: NCT05776823
Title: Pharmacist-Led Interventions to Increase Access to Medications for Opioid Use Disorder
Brief Title: Pharmacist-Led Interventions to Increase Access to Medications for Opioid Use Disorders (PLI-MOUD)
Acronym: PLI-MOUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 274818
Record Dates: First submitted 2023-03-01; First posted 2023-03-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder; Overdose
Keywords: Harm Reduction; Criminal Justice; Pharmacy Practice
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose; Harm Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pharmacist Narcan Training (Experimental): Pharmacist-led intervention
  Interventions: Behavioral: Pharmacist Narcan Training
- Substance Use Counselor Narcan Training (Active Comparator): Non-clinician intervention
  Interventions: Behavioral: Substance Use Counselor Narcan Training
- Brief Intervention and Referral to Treatment (BIRT) (Experimental): BIRT intervention
  Interventions: Behavioral: BIRT
- Standard Medication Counseling (SMC) (Active Comparator): SMC intervention
  Interventions: Behavioral: SMC

INTERVENTIONS:
Behavioral: Pharmacist Narcan Training — A 20-45-minute didactic presentation conducted with a skills training component designed to demonstrate appropriate administration of the Narcan nasal spray.
  Arms: Pharmacist Narcan Training
Behavioral: BIRT — BIRT participants will receive a 30-45-minute session delivered by the pharmacist to introduce and encourage treatment options, MOUD information, OUD information, and treatment facility information (i.e., flyers (RDD study/CAST clinic/State Opioid Response III funded agencies) and educational materials), and a referral to treatment/linkage to service providers.
  Arms: Brief Intervention and Referral to Treatment (BIRT)
Behavioral: SMC — SMS participants will receive a 5-10-minute counseling session delivered by the pharmacist providing MOUD information, OUD information, and treatment facility information (i.e., flyers (RDD study/CAST clinic/State Opioid Response III funded agencies) and educational materials).
  Arms: Standard Medication Counseling (SMC)
Behavioral: Substance Use Counselor Narcan Training — A 20-45-minute didactic presentation conducted with a skills training component designed to demonstrate appropriate administration of the Narcan nasal spray.
  Arms: Substance Use Counselor Narcan Training

SUMMARY:
The purpose of this study is to investigate the impact of a pharmacist-led intervention to expand access to medications for opioid use disorder (MOUD) on racial/ethnic differences in opioid-related overdose among individuals diagnosed with opioid use disorder (OUD) currently incarcerated in a carceral setting. In this study, participants will be screened for opioid use, trained to administer Narcan nasal spray, receive motivational counseling and referral to treatment post-release from a carceral setting (a Re-Entry program) into the community.

DETAILED DESCRIPTION:
The main objectives of this study are:

1. To increase understanding of racial/ethnic differences in the prevalence of OUD.
2. To test if a pharmacist-led intervention is more effective than a substance use counselor (lay person) in increasing knowledge and confidence among different racial/ethnic groups related to administering Narcan nasal spray in an opioid overdose situation.
3. To test if a pharmacist-delivered an evidence-based intervention, q brief intervention and referral to treatment (BIRT) versus standard medication counseling (SMC) is more effective in increasing access to MOUD.

ELIGIBILITY:
Inclusion Criteria

Narcan Training:

* a Re-Entry program participant 7-14 days from release from carceral setting
* provide collateral contact information for ≥2 persons (to ensure consistent contact/follow up)
* have a reliable landline or mobile phone to be contacted by pharmacist
* plan to remain in the Little Rock area for at least 6 months
* able to read and write English
* able to provide informed consent
* possesses manual dexterity; physical ability to roll a person onto her/his/their back and side
* have no allergy to naloxone hydrochloride (active ingredient in Narcan nasal spray)-
* identified on the RODS screener as positive for OUD.

BIRT/SMC:

* a Re-Entry program participant 7-14 days from release from the carceral setting
* provide contact information for ≥2 persons (to ensure consistent contact/follow -up)
* have a reliable landline or mobile phone to be contacted by pharmacist
* plan to remain in the Little Rock area for at least 6 months
* able to read and write English; able to provide informed consent
* identified with OUD.

Exclusion Criteria:

Narcan training:

* not a RE-entry program participant
* identified substance use disorders other than OUD

BIRT/SMC:

* not a RE-entry program participant
* identified substance use disorders other than OUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Opioid overdose training | at month 6
  Participants' knowledge about opioid overdose and confidence to recognize and respond to opioid overdose situations as a function of the trainer. Participants will complete a brief validated survey, the adapted Perceived Competence Scale. The questions on the survey are rated on a 7-point scale and participants indicate how true four statements are about their ability to recognize and respond to overdoses: the scale, 1 (not at all true) to 7 (very true).
Retention | at month 6
  Participants, regardless of treatment arm, will receive follow-up telephone interviews at 6 months post-release from the carceral setting into the community. Interviews will address the primary question whether MOUD treatment was initiated and maintained.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan N Breckling, PharmD, Principal Investigator — UAMS
Locations (1):
- Pulaski County Regional Detention Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No